CLINICAL TRIAL: NCT07382258
Title: A Prospective, Single-Center Study of Inhaled Nitric Oxide in Individuals Diagnosed With Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Study of Inhaled Nitric Oxide in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novlead Inc. (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-COPD
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iNO 10 ppm Dose Group (Experimental): Participants will receive inhaled nitric oxide at a concentration of 10 ppm, for a minimum of 2 hours per day, over 7 consecutive days.
  Interventions: Device: Nitric Oxide Generation and Delivery System
- iNO 40 ppm Dose Group (Experimental): Participants will receive inhaled nitric oxide at a concentration of 40 ppm, for a minimum of 2 hours per day, over 7 consecutive days.
  Interventions: Device: Nitric Oxide Generation and Delivery System

INTERVENTIONS:
Device: Nitric Oxide Generation and Delivery System — A device designed to deliver a stable, user-prescribed concentration of nitric oxide gas into the inspiratory circuit of the patient's breathing apparatus for inhalation therapy.

SUMMARY:
This clinical trial aims to assess the impact on exercise tolerance and the safety of inhaled nitric oxide in subjects with moderate-to-severe COPD. The findings are expected to contribute to the development of safe and effective therapeutic strategies for COPD management.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40 and 75 years, inclusive.
2. History of smoking with a cumulative exposure of ≥10 pack-years, and having ceased smoking for at least one month prior to study participation.
3. Diagnosis of moderate-to-severe COPD confirmed by post-bronchodilator spirometry: FEV1/FVC < 0.7 and FEV1 between 30% and 80% of predicted value.
4. Willing and able to provide written informed consent and comply with all study-related procedures.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Use of nicotine-containing products (e.g., patches, gum) within the past month.
3. Current diagnosis of asthma or any other active respiratory condition considered non-COPD by the investigator.
4. Physical obstruction of the nasal passages.
5. Experienced a COPD exacerbation within the past month requiring initiation or escalation of systemic corticosteroids.
6. Impaired left ventricular systolic function, defined as left ventricular ejection fraction (LVEF) < 50%.
7. Significant valvular heart disease (moderate/severe aortic or mitral stenosis/regurgitation) or prior mitral valve replacement.
8. Use of approved pulmonary hypertension medications (e.g., sildenafil, bosentan, prostacyclins) within 30 days prior to screening or during the study.
9. Participation in another interventional clinical trial involving drugs or devices within 30 days prior to enrollment.
10. Any other medical or psychiatric condition that, in the investigator's judgment, would compromise patient safety or study integrity.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Oxygen Uptake (VO2max) | Baseline, Day 7
  The difference in VO2max values measured during cardiopulmonary exercise testing before and after the one-week iNO treatment period.
Change in Ventilatory Efficiency (VE/VCO2) | Baseline, Day 7
  The difference in the minute ventilation-to-carbon dioxide output (VE/VCO2) ratio measured during cardiopulmonary exercise testing before and after the one-week iNO treatment period.
Change in Oxygen Uptake to Work Rate Ratio (ΔVO2/ΔW) | Baseline, Day 7
  The difference in the ratio of change in oxygen uptake to change in work rate (ΔVO2/ΔW) measured during cardiopulmonary exercise testing before and after the one-week iNO treatment period.
Change in Perceived Exertion (Borg Score) | Baseline, Day 7
  The difference in Borg scale scores for perceived exertion recorded during cardiopulmonary exercise testing before and after the one-week iNO treatment period.

SECONDARY OUTCOMES:
Change in COPD Assessment Test (CAT) Score | Baseline, Day 7
  The difference in total CAT score (range 0-40, higher scores indicate worse health status) reported before and after the one-week iNO treatment period.
Change in Modified Medical Research Council (mMRC) Dyspnea Scale Score | Baseline, Day 7
  The difference in mMRC dyspnea scale score (range 0-4, higher scores indicate greater breathlessness) reported before and after the one-week iNO treatment period.
Change in Six-Minute Walk Distance (6MWD) | Baseline, Day 7
  The difference in the distance walked during a six-minute walk test performed before and after the one-week iNO treatment period.
Change in Forced Expiratory Volume in 1 Second (FEV1) | Baseline, Day 7
  The difference in FEV1 values from pulmonary function tests performed before and after the one-week iNO treatment period.
Change in Forced Vital Capacity (FVC) | Baseline, Day 7
  The difference in FVC values from pulmonary function tests performed before and after the one-week iNO treatment period.
Change in FEV1/FVC Ratio | Baseline, Day 7
  The difference in the FEV1/FVC ratio from pulmonary function tests performed before and after the one-week iNO treatment period.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline up to Day 7
  Proportion of participants experiencing any adverse event during the treatment period, calculated as (Number of subjects with adverse events / Total number of treated subjects) * 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No